CLINICAL TRIAL: NCT02981875
Title: Oculomotor Training Improves Reading Eye Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Carly Lam, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HongKongPUVT
Record Dates: First submitted 2016-08-17; First posted 2016-12-05 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Ocular Motility Disorders
Keywords: reading eye movement
MeSH Terms: conditions — Ocular Motility Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental (Experimental): oculomotor training
  Interventions: Other: oculomotor training
- control (Placebo Comparator): placebo vision training exercises
  Interventions: Other: placebo

INTERVENTIONS:
Other: oculomotor training — a sequence of vision training exercises which focused mainly in oculomotor skill
  Arms: experimental
Other: placebo — placebo vision training exercises involving minimal accommodation and vergence eye movement.
  Arms: control

SUMMARY:
Children with reading eye movement problems were recruited for this study. The treatment group was provided with oculomotor training for 8 weeks, the control group was given placebo exercises.

DETAILED DESCRIPTION:
Purpose of study Reading is one of the integral elements for learning and poor readers were reported to have less efficient reading eye movements. They were typically characterized by having higher number in fixation and regression, reduced reading speed and perceptual span. The purpose of this study was to investigate if vision therapy which limited to training of oculomotor skills can improve reading eye movement.

Methodology This was a randomized, prospective study. 30 subjects aged from 8-9 years of age with reading difficulties and reading eye movement problems were recruited. They all have normal intelligence and ocular health, but failed to meet the Taylor reading eye movement norms when tested with the Visagraph III. The subjects were randomly assigned into either the treatment group (15) or the control group (15). The treatment group had to go through a course of oculomotor vision therapy and the control group was given placebo exercises. Vision therapy for the treatment group involved 8 weeks of training (office training - 3 times a week, 30 min per session; home training - 4 times a week, 30 min per session). Office training involved the use of Vis-Flex (Visual Flexibility Trainer - an electronic device with L.E.D. lights which can display various flashing patterns at variable speeds). Home training involved several saccadic eye movement exercises. Subjects and parents were also asked to grade the reading symptoms checklist before and after the training.

ELIGIBILITY:
Inclusion Criteria:

* Reported by teachers or parents to have reading difficulties and failed to meet the Taylor reading eye movement norms when tested with the Visagraph III (below age norm for both fixation and regression number).
* Studying in mainstream primary schools (8-9 years of age)
* With normal near visual acuities for both eyes (with or without spectacles)
* Hyperopia below +4.00 D
* Myopia below -4.00 D
* Astigmatism below -2.00 D
* Anisometropia less than 2.0 D difference between the two eyes
* Near heterophoria within 0-4 exophoria
* Vertical heterophoria less than 1 prism dioptre
* Monocular amplitude of accommodation over 10 D in both eyes
* With parents who were willing to perform vision therapy exercises for the children at home on a regular basis
* Both genders were acceptable as Eden et al (1994) stated that gender had no effect on oculomotor skills

Exclusion criteria:

* With strabismus
* Presence of eye diseases
* History of dyslexia (learning disability) or developmental delay

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in number of fixation and regression during reading after 8 weeks of oculomotor training | 8 weeks
  number of fixation and regression is measured by Visagraph per 100 words

SECONDARY OUTCOMES:
Change in reading rate during reading after 8 weeks of oculomotor training | 8 weeks
  reading rate in number of words/min and fixation duration measured in seconds
Change in perceptual span (words per fixation) during reading after 8 weeks of oculomotor training | 8 weeks
  perceptual span measured in words per fixation
Change in fixation duration (seconds) during reading after 8 weeks of oculomotor training | 8 weeks
  fixation duration measured in seconds
Change in symptom scores after 8 weeks of oculomotor training | 8 weeks
  symptom scores is calculated with a scale of 0 to 4 for all the 8 items of manifested symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Carly SY Lam, Principal Investigator — The Hong Kong Polytechnic University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bigelow ER, McKenzie BE. Unstable ocular dominance and reading ability. Perception. 1985;14(3):329-35. doi: 10.1068/p140329. PMID 4088794
- [Background] Biscaldi M, Gezeck S, Stuhr V. Poor saccadic control correlates with dyslexia. Neuropsychologia. 1998 Nov;36(11):1189-202. doi: 10.1016/s0028-3932(97)00170-x. PMID 9842764
- [Background] Borsting EJ, Rouse MW, Mitchell GL, Scheiman M, Cotter SA, Cooper J, Kulp MT, London R; Convergence Insufficiency Treatment Trial Group. Validity and reliability of the revised convergence insufficiency symptom survey in children aged 9 to 18 years. Optom Vis Sci. 2003 Dec;80(12):832-8. doi: 10.1097/00006324-200312000-00014. PMID 14688547
- [Background] Bosse ML, Tainturier MJ, Valdois S. Developmental dyslexia: the visual attention span deficit hypothesis. Cognition. 2007 Aug;104(2):198-230. doi: 10.1016/j.cognition.2006.05.009. Epub 2006 Jul 21. PMID 16859667
- [Background] Bucci MP, Nassibi N, Gerard CL, Bui-Quoc E, Seassau M. Immaturity of the oculomotor saccade and vergence interaction in dyslexic children: evidence from a reading and visual search study. PLoS One. 2012;7(3):e33458. doi: 10.1371/journal.pone.0033458. Epub 2012 Mar 16. PMID 22438934
- [Background] Eden GF, Stein JF, Wood HM, Wood FB. Differences in eye movements and reading problems in dyslexic and normal children. Vision Res. 1994 May;34(10):1345-58. doi: 10.1016/0042-6989(94)90209-7. PMID 8023443
- [Background] Hutzler F, Wimmer H. Eye movements of dyslexic children when reading in a regular orthography. Brain Lang. 2004 Apr;89(1):235-42. doi: 10.1016/S0093-934X(03)00401-2. PMID 15010255
- [Background] Jainta S, Kapoula Z. Dyslexic children are confronted with unstable binocular fixation while reading. PLoS One. 2011 Apr 6;6(4):e18694. doi: 10.1371/journal.pone.0018694. PMID 21494641
- [Background] McConkie GW, Kerr PW, Reddix MD, Zola D. Eye movement control during reading: I. The location of initial eye fixations on words. Vision Res. 1988;28(10):1107-18. doi: 10.1016/0042-6989(88)90137-x. PMID 3257013
- [Background] McConkie GW, Kerr PW, Reddix MD, Zola D, Jacobs AM. Eye movement control during reading: II. Frequency of refixating a word. Percept Psychophys. 1989 Sep;46(3):245-53. doi: 10.3758/bf03208086. PMID 2771616
- [Background] Pavlidis GT. Eye movement differences between dyslexics, normal, and retarded readers while sequentially fixating digits. Am J Optom Physiol Opt. 1985 Dec;62(12):820-32. doi: 10.1097/00006324-198512000-00003. PMID 4083326
- [Background] Poynter HL, Schor C, Haynes HM, Hirsch J. Oculomotor functions in reading disability. Am J Optom Physiol Opt. 1982 Feb;59(2):116-27. doi: 10.1097/00006324-198202000-00002. PMID 7065104
- [Background] Prado C, Dubois M, Valdois S. The eye movements of dyslexic children during reading and visual search: impact of the visual attention span. Vision Res. 2007 Sep;47(19):2521-30. doi: 10.1016/j.visres.2007.06.001. Epub 2007 Aug 23. PMID 17719073
- [Background] Rounds BB, Manley CW, Norris RH. The effect of oculomotor training on reading efficiency. J Am Optom Assoc. 1991 Feb;62(2):92-9. PMID 1814996
- [Background] Shainberg MJ. Vision therapy and orthoptics. Am Orthopt J. 2010;60:28-32. doi: 10.3368/aoj.60.1.28. PMID 21061881
- [Background] Solan HA. Deficient eye-movement patterns in achieving high school students: three case histories. J Learn Disabil. 1985 Feb;18(2):66-70. doi: 10.1177/002221948501800201. No abstract available. PMID 3973502
- [Background] Solan HA. Eye movement problems in achieving readers: an update. Am J Optom Physiol Opt. 1985 Dec;62(12):812-9. doi: 10.1097/00006324-198512000-00002. PMID 4083325